CLINICAL TRIAL: NCT05526196
Title: Combined and Separate Effects of Cannabis and Tobacco: Psychomotor, Subjective and Physiological Outcomes
Acronym: CASE-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 130-2021
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Driving Under the Influence
MeSH Terms: conditions — Driving Under the Influence | interventions — nabiximols; Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Other): A cigarette containing placebo cannabis and placebo tobacco
  Interventions: Drug: Placebo
- Tobacco (Other): A cigarette with placebo cannabis and active tobacco
  Interventions: Drug: Tobacco
- Cannabis (Other): A cigarette with active cannabis and placebo tobacco
  Interventions: Drug: Cannabis
- Tobacco and cannabis (Other): A cigarette with active cannabis and active tobacco
  Interventions: Drug: Cannabis tobacco

INTERVENTIONS:
Drug: Cannabis — Dried flower cannabis cigarette with 22% THC
  Arms: Cannabis
Drug: Tobacco — Dried flower cigarette with active nicotine
  Arms: Tobacco
Drug: Cannabis tobacco — Dried flower cigarette with active nicotine and cannabis
  Arms: Tobacco and cannabis
Drug: Placebo — Dried flower cigarette with both placebo tobacco and cannabis
  Arms: Placebo

SUMMARY:
Co-administration of cannabis and tobacco is a common practice, but there is little experimental evidence aimed at understanding the reasons for this prevalence. Some preliminary evidence suggests that tobacco may actually counteract the cognitive-impairing effects of cannabis, and may also increase the subjective ('liking') effects of cannabis, but results are inconclusive. Further, there are no studies into the effects of tobacco on other cannabis-related harms such as driving, or on the ability of tobacco to alter the blood levels of THC, the chemical responsible for the psychoactive properties of cannabis. The purpose of the present study will be to evaluate the effects of tobacco, cannabis or combinations of tobacco and cannabis on driving, cognition, subjective effects and blood THC. Driving will be assessed using a state-of-the-art driving simulator that allows for the safe and objective measurement of the effects of intoxicating substances on driving. Participants will be regular users of cannabis and will be invited to the lab for four counterbalanced test sessions. In these test sessions they will drive the simulator and undergo cognitive tests before and after smoking: 1) cannabis; 2) tobacco; 3) cannabis + tobacco; or 4) placebo. Outcomes will be measured at several time points after smoking the product. Participants will also give blood for determination of levels of THC, and will complete subjective effects questionnaires both before and after smoking the cigarette. This study will be one of the first experimental laboratory studies of the reasons behind co-administration of tobacco and cannabis.

ELIGIBILITY:
Inclusion Criteria:

* • Adults aged 19 years to 45 years (to control for the effects of age on cognition)

  * Smoke or vape cannabis at least once a month but no more than 4 times a week (to avoid enrolling people with cannabis use disorder who may experience withdrawal when asked to abstain from cannabis)
  * Experience with smoked cannabis in the past year
  * Report use of at least 100 cigarettes in their lifetime to ensure familiarity with the tobacco used in the present study
  * Use of any nicotine (smoked, vaped, etc) in the past year
  * G2 or full G driver's licence for at least a year
  * Willing to abstain from alcohol and other drugs (other than drugs required for treatment of a medical condition) for 48 hours prior to study session
  * Normal heart rate and blood pressure as determined by the QI (because cannabis and tobacco increase heart rate)
  * Normal ECG (because cannabis and tobacco increase heart rate)
  * Willing to abstain from cannabis for 72 hours prior to the test session and from smoking tobacco for 12 hours
  * Willing to use an accepted form of contraception during the study (both males and females)
  * Past lifetime experience with co-use of cannabis or tobacco (either simultaneous or concurrent)
  * Provides written and informed consent

Exclusion Criteria:

* • Use of psychoactive medications or drugs

  * Current alcohol or other substance use disorder, including cannabis (as assessed with the SCID)
  * Current or past nicotine dependence (to avoid precipitating a relapse)
  * Withdrawal symptoms as assessed with the Marijuana Withdrawal Checklist [57, 58]
  * A score of less than 10 on the Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) [59]
  * Family history of schizophrenia or psychosis (to avoid giving cannabis to anyone with a predisposition to psychosis)
  * Respiratory illnesses (due to the smoked route of administration in this study)
  * Any serious medical condition precluding participation as judged by the responsible study physician
  * Pregnancy or breastfeeding
  * Negative urine screen for cannabis at eligibility assessment (to ensure experience with cannabis)
  * Neurological disorders that may affect cognitive function
  * Treatment-seeking for tobacco or cannabis use
  * Use of more than 5 cigarettes a day (to avoid confound of the effects of chronic smoking on measures)
  * Concomitant therapy with sedative-hypnotics or other psychoactive drugs (counter-indicated with cannabis)

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Standard deviation of lateral position | baseline
  car 'weaving'
Standard deviation of lateral position | 15 minutes post smoking
  car 'weaving'
Standard deviation of lateral position | 180 minutes post smoking
  car 'weaving'

SECONDARY OUTCOMES:
Speed | baseline
  Speed (in km) of the car
Speed | 15 minutes post smoking
  Speed (in km) of the car
Speed | 180 minutes post smoking
  Speed (in km) of the car
Reaction time | baseline
  Time to hit the brake after introduction of an obstacle
Reaction time | 15 minutes post smoking
  Time to hit the brake after introduction of an obstacle
Reaction time | 180 minutes post smoking
  Time to hit the brake after introduction of an obstacle
Collisions | baseline
  number of times the car hit an obstacle
Collisions | 15 minutes post smoking
  number of times the car hit an obstacle
Collisions | 180 minutes post smoking
  number of times the car hit an obstacle
Concentration of THC (ng/ml) | Baseline
  Psychoactive component of cannabis
Concentration of THC (ng/ml) | 15 minutes post smoking
  Psychoactive component of cannabis
Useful Field of View Processing Speed | baseline
  Mean threshold for discriminating stimuli presented in central vision
Useful Field of View Processing Speed | 60 minutes post smoking
  Mean threshold for discriminating stimuli presented in central vision
Useful Field of View Processing Speed | 210 minutes post smoking
  Mean threshold for discriminating stimuli presented in central vision
Useful Field of View Divided attention | baseline
  Mean threshold for discriminating stimuli presented in central vision, with a concurrent perpheral target task
Useful Field of View Divided attention | 60 minutes
  Mean threshold for discriminating stimuli presented in central vision, with a concurrent perpheral target task
Useful Field of View Divided attention | 210 minutes
  Mean threshold for discriminating stimuli presented in central vision, with a concurrent perpheral target task
Useful Field of View Selective attention | baseline
  Mean threshold for divided attention but with distractors
Useful Field of View Selective attention | 60 minutes
  Mean threshold for divided attention but with distractors
Useful Field of View Selective attention | 210 minutes
  Mean threshold for divided attention but with distractors
Trail making task | baseline
  Cognitive assessment
Trail making task | 60 minutes post smoking
  Cognitive assessment
Trail making task | 210 minutes post smoking
  Cognitive assessment
Verbal free recall | baseline
  Test of memory
Verbal free recall | 60 minutes post smoking
  Test of memory
Verbal free recall | 210 minutes post smoking
  Test of memory
Addiction Research Centre Inventory | baseline
  Test of mood with 53 true-false questions that are summed to produce a measure of the intensity of mood, with higher scores reflecting greater mood
Addiction Research Centre Inventory | 60 minutes post smoking
  Test of mood with 53 true-false questions that are summed to produce a measure of the intensity of mood, with higher scores reflecting greater mood
Addiction Research Centre Inventory | 210 minutes post smoking
  Test of mood with 53 true-false questions that are summed to produce a measure of the intensity of mood, with higher scores reflecting greater mood
Profile of Mood States | baseline
  Test of mood with 76 items with a five point scale that are summed to produce a measure of the intensity of mood, with higher scores indicating more agreemen
Profile of Mood States | 60 minutes post smoking
  Test of mood with 76 items with a five point scale that are summed to produce a measure of the intensity of mood, with higher scores indicating more agreemen
Profile of Mood States | 210 minutes post smoking
  Test of mood with 76 items with a five point scale that are summed to produce a measure of the intensity of mood, with higher scores indicating more agreemen
Visual Analog Scale | baseline
  test of mood on a scale from 0 to 100, with greater number indicating more agreement
Visual Analog Scale | 15 minutes post smoking
  test of mood on a scale from 0 to 100, with greater number indicating more agreement
Visual Analog Scale | 60 minutes post smoking
  test of mood on a scale from 0 to 100, with greater number indicating more agreement
Visual Analog Scale | 120 minutes post smoking
  test of mood on a scale from 0 to 100, with greater number indicating more agreement
Visual Analog Scale | 180 minutes post smoking
  test of mood on a scale from 0 to 100, with greater number indicating more agreement
Visual Analog Scale | 240 minutes post smoking
  test of mood on a scale from 0 to 100, with greater number indicating more agreement
Visual Analog Scale | 300 minutes post smoking
  test of mood on a scale from 0 to 100, with greater number indicating more agreement

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No